CLINICAL TRIAL: NCT04331041
Title: Phase II Study of Stereotactic Body Radiotherapy and Focal Adhesion Kinase Inhibitor in Advanced Pancreas Adenocarcinoma
Brief Title: Stereotactic Body Radiotherapy and Focal Adhesion Kinase Inhibitor in Advanced Pancreas Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202106061; R01CA248917-01 (NIH)
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Pancreas Cancer; Cancer of the Pancreas; Pancreas Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — defactinib

STUDY DESIGN:
Intervention Model Description: The enrolled patients are 6:1 randomized to either Experimental Arm or Adaptive Comparator Arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Adaptive SBRT + Defactinib (Experimental): * Participants in this study will receive 5 fractions of magnetic resonance adaptive stereotactic body radiation therapy (SBRT) and seventeen 21-day cycles of defactinib (beginning on Day 2 of radiation).
  * Participants who are candidates for surgical resection will undergo standard of care surgery at 2 weeks post-end of SBRT (+/- 1 weeks) or 12 weeks post-end of SBRT (+/- 1 week). These participants will discontinue defactinib the day prior to the operation and will resume taking it for the remainder of the 17 cycles 4 to 6 weeks after surgery. Participants who are not candidates for surgical resection will continue to receive defactinib uninterrupted. All participants should receive 17 cycles of defactinib unless they experience disease progression or intolerable toxicity.
  Interventions: Device: Adaptive stereotactic body radiation therapy; Drug: Defactinib; Procedure: Tumor biopsy; Procedure: Research blood draw
- Adaptive SBRT (Active Comparator): -Participants in this study will receive 5 fractions of magnetic resonance adaptive stereotactic body radiation therapy (SBRT)
  Interventions: Device: Adaptive stereotactic body radiation therapy; Procedure: Research blood draw

INTERVENTIONS:
Device: Adaptive stereotactic body radiation therapy — * Will be administered using MRIdian and Ethos
  * 50 Gy in 5 fractions
  Other Names: Adaptive SBRT
Drug: Defactinib — -Oral drug 400 mg twice a day
  Other Names: VS-6063; PF-04554878
  Arms: Adaptive SBRT + Defactinib
Procedure: Tumor biopsy — -Baseline and 12-14 weeks after end of SBRT (or at time of surgery)
  Arms: Adaptive SBRT + Defactinib
Procedure: Research blood draw — -Baseline, 6-8 weeks after the end of SBRT, and 12-14 weeks after the end of SBRT

SUMMARY:
Patients with advanced pancreas adenocarcinoma will be randomized on a 6:1 basis to receive standard of care chemotherapy followed by adaptive stereotactic body radiotherapy (SBRT) with concurrent and adjuvant FAK inhibitor defactinib (experimental arm) or standard of care chemotherapy followed by SBRT (control arm). Patients enrolled to the experimental arm will be assessed for clinical outcomes such as progression free survival (PFS), local control, distant control, and toxicity. The initial 6 patients randomized to the experimental arm will be considered the safety lead-in and will be assessed for dose-limiting toxicities (DLTs). Following completion of the safety lead-in, additional patients will be accrued in order to reach a total of 36 patients on the experimental arm (inclusive of the safety lead-in cohort) and 6 on the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced pancreas adenocarcinoma that is considered borderline resectable or unresectable per institutional standardized criteria of unresectability or medical inoperability (NCCN guidelines 2.2021 PANC-C 1 of 2).
* Patients with locoregional adenopathy are eligible as long as all suspicious lymph nodes are deemed to be adjacent to the primary tumor as per radiation oncologist assessment.
* At least 3 months of systemic chemotherapy for this disease without progression of local or systemic disease. Newly diagnosed patients may be screened for enrollment in this study and can be enrolled once they have completed 3 months of systemic chemotherapy (and still meet all eligibility criteria) prior to the start of study treatment.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Life expectancy > 3 months
* Normal bone marrow and organ function within 21 days of randomization as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN; no prior history of Gilbert's syndrome
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN or ≤ 5.0 x IULN if due to liver involvement by tumor
  * Creatinine clearance ≤ 1.5 x IULN or glomerular filtration rate of ≥ 60 mL/min
  * INR ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
  * aPTT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as INR or PTT is within therapeutic range of intended use of anticoagulants
  * Albumin ≥ 2.5 mg/dL
* Corrected QT interval (QTc) < 480 ms (as calculated by the Fridericia correction formula).
* The effects of defactinib on the developing human fetus are unknown. For this reason and because radiation therapy is known to be teratogenic, women of childbearing potential and men must agree to use highly effective contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and 120 days after completion of the study
* Ability to understand and willingness to sign an IRB approved written informed consent document

Exclusion Criteria:

* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease.
* Clinical evident ascites or pleural effusion that requires therapeutic paracentesis or thoracentesis.
* Prior treatment with a drug of the FAK inhibitor class or with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte associated antigen 4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Prior anti-human antibody response (AHA or ADA).
* Currently receiving any other investigational agents or has receive any other investigational agents within 4 weeks or 5 half-lives or planned first dose of study agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to defactinib or other agents used in the study.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy not routinely associated with chemotherapeutic regimen.
* Requires continued use of warfarin for anticoagulation and cannot stop warfarin or be safely switched to another anticoagulant or direct oral anticoagulant
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, hypertension, immunosuppression, autoimmune conditions, or underlying pulmonary disease.
* Has an active autoimmune disease requiring systemic treatment within the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Received a live vaccine within 30 days prior to the first study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed.
* Known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV RNA [qualitative] is detected).
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has a known history of active TB (bacillus tuberculosis).
* Major surgery within 28 days prior to the first study treatment.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.
* Known SARS-Cov2 infection ≤28 days prior to first dose of study therapy.
* Exposure to P-glycoprotein (P-gp) inhibitors or inducers within 14 days prior to the first dose and during the course of therapy.
* Subjects with the inability to swallow oral medications or impaired gastrointestinal absorption due to gastrectomy or active inflammatory bowel disease.
* Subjects with a history of hypersensitivity to any of the inactive ingredients (hydroxypropylmethylcellulose, mannitol, magnesium stearate) of the investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) (Experimental Arm only) | After completion of treatment (estimated to be 12 months)
  * PFS is defined as the duration of time from start of standard of care chemotherapy treatment to time of progression or death, whichever occurs first. The alive patients without progression will be censored at the last follow-up.
  * Progressive disease: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).

SECONDARY OUTCOMES:
Number of participants with acute adverse events (Experimental Arm only) | From start of adaptive SBRT through 90 days
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Number of participants with late adverse events (Experimental Arm only) | From 91 days through completion of follow-up (estimated to be 24 months)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Overall survival (Experimental Arm only) | Through completion of follow-up (estimated to be 24 months)
  -Overall survival as defined as the time from the date of treatment until death; censored at last follow-up if death is not observed
Distant metastasis progression-free survival (DM-PFS) (Experimental Arm only) | Through completion of follow-up (estimated to be 24 months)
  -Defined as the days from the date of the treatment to distant metastasis progression or death
Objective response rate (Experimental Arm only) | 12-14 weeks post-adaptive SBRT
  -Objective response rate as determined by RECIST 1.1 criteria, with one change. Patients who undergo resection will be considered to have a CR if there is a pathologic complete response (pCR) on the surgical specimen. After resection, patients will no longer be evaluated for ORR.
Local control (Experimental Arm only) | Through completion of follow-up (estimated to be 24 months)
  -Local control as defined by no progression of the primary tumor by RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Carl DeSelm, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of individual participant data that underlie the results reported in the article after deidentification (text, tables, figures, and appendices) for individual participant data meta-analysis.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators who proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Derived] Fard D, Giraudo E, Tamagnone L. Mind the (guidance) signals! Translational relevance of semaphorins, plexins, and neuropilins in pancreatic cancer. Trends Mol Med. 2023 Oct;29(10):817-829. doi: 10.1016/j.molmed.2023.07.009. Epub 2023 Aug 17. PMID 37598000
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu